CLINICAL TRIAL: NCT00215163
Title: Randomized Trial of Paroxetine-CR for the Treatment of Patients With Post-Traumatic Stress Disorder (PTSD) Remaining Symptomatic After Initial Exposure Therapy
Brief Title: Paroxetine-CR to Treat Post-Traumatic Stress Disorder (PTSD) Symptomatic After Initial Exposure Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4304; 4304-02-12 (Other: Duke IRB#)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Anxiety; CBT; Exposure; Paroxetine; Paroxetine-CR
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Cognitive-behavioral therapy and paroxetine-CR

SUMMARY:
Both pharmacotherapeutic and psychosocial interventions have domenstrated efficacy for PTSD. However, although these interventions can be helpful, many patients remain symptomatic despite initial treatment. In this study, we will examine the relative efficacy of the addition of paroxetine-CR compared to placebo for patients remaining symptomatic despite a brief and intensive course of cognitive-behavioral therapy (CBT).

DETAILED DESCRIPTION:
This is a systematic controlled study examining the use of augmentation with pharmaotherapy for PTSD patients remaining symptomatic despite CBT (exposure therapy). The aims of the study include examination of: (1) the efficacy of paroxetine-CR compared to placebo as additions to ongoing exposure therapy in patients who failed to respond to brief, intensive CBT; (2) the tolerability of paroxetine-CR compared to placebo as additions to ongoing exposure therapy in patients who failed to respond to brief, intensive CBT; (3) the outcome of patients at 6 months follow-up to randomized treatment. Patients will initially have intensive (8 sessions over 4 weeks) prolonged exposure therapy. Patients who remain symptomatic will be randomzied to receive either flexibly-dosed paroxetine-CR (12.5 mg/d - 62.5 mg/d) or placebo in conjunction with additional 5 sessions of prolonged exposure over 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age with a primary (the condition that is most central to the patient's current distress) psychiatric diagnosis of PTSD as defined by DSM-IV criteria
* Patients must have remained symptomatic (CGI-S > or = 3) and a score of at least 6 on the SPRINT after a minimum of 7 sessions of prolonged exposure (delivered within 6 weeks) to be eligible for randomized treatment.

Exclusion Criteria:

* Serious medical illness or instability for which hospitalization may be likely within the next 3 months
* Pregnant or lactating women or those of childbearing potential not using medically accepted forms of contraception
* Concurrent use of other psychotropic medications
* Lifetime diagnosis of schizophrenia or any other psychotic disorder, mental retardation, organic mental disorders, or bipolar disorder
* Obsessive-Compulsive Disorder, eating disorders, or alcohol/substance abuse disorders within the last 6 months
* A current primary diagnosis of major depression, dysthymia, social anxiety disorder, and generalized anxiety disorder
* A history of hypersensitivity or poor response to paroxetine or those using antidepressants, buspirone, or beta-blockers within 2 weeks of randomization
* Concurrent dynamic or supportive psychotherapy if started within 2 months prior to onset of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-12; Study Completion 2006-06

PRIMARY OUTCOMES:
Short PTSD Rating Interview (SPRINT)
Davidson Trauma Scale (DTS)

SECONDARY OUTCOMES:
Clinical Global Impressions Severity Scale (CGI-S)
Clinical Global Impressions Improvement Scale (CGI-I)
Posttraumatic Diagnostic Scale (PDS)
Beck Depression Inventory (BDI)
Quality of Life Enjoyment and Satisfaction Questionnaire/General Activities Subscale (Q-LES-Q/GA)
Sheehan Disability Scale (SDS)
Connor-Davidson Resilience Scale (CD-RISC)
Post-Traumatic Cognitions Inventory (PTCI)
Severity of Symptoms Scale (SOSS)
Pittsburgh Sleep Quality Index (PSQI)
World Assumptions Scale (WAS)
Mood-SR Lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, M.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of California at San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Simon NM, Connor KM, Lang AJ, Rauch S, Krulewicz S, LeBeau RT, Davidson JR, Stein MB, Otto MW, Foa EB, Pollack MH. Paroxetine CR augmentation for posttraumatic stress disorder refractory to prolonged exposure therapy. J Clin Psychiatry. 2008 Mar;69(3):400-5. doi: 10.4088/jcp.v69n0309. PMID 18348595